CLINICAL TRIAL: NCT05063344
Title: NOWDx Test for the Diagnosis of Syphilis
Status: Completed | Type: Observational
Sponsor: NOWDiagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NOWDx Syphilis Study
Record Dates: First submitted 2020-03-01; First posted 2021-10-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Syphilis Infection; Treponema Pallidum Infection
Keywords: Syphilis; Treponema Pallidum
MeSH Terms: conditions — Syphilis; Treponemal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Sexually active persons who self-select for syphilis testing: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years
  Interventions: Device: Diagnostic Test: NOWDx Syphilis Test
- Expectant mothers: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years
  Interventions: Device: Diagnostic Test: NOWDx Syphilis Test
- Lay users: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years; 1/2 high risk sexual behavior and 1/2 low risk sexual behavior
  Interventions: Device: Diagnostic Test: NOWDx Syphilis Test

INTERVENTIONS:
Device: Diagnostic Test: NOWDx Syphilis Test — For this observational trial, the Intervention of interest is the NOWDx Syphilis Test.

SUMMARY:
This study is designed to compare the performance of the NOWDx Syphilis Test to a currently marketed device. The intent is to show the rapid test device is comparable to the currently marketed device. The NOWDx Syphilis Test is intended for qualitatively detecting the presence or absence of human antibodies to syphilis in human whole blood to aid in the diagnosis of infection caused by Treponema pallidum.

DETAILED DESCRIPTION:
The objective of this study is to establish the performance characteristics of the NOWDx Syphilis Test based on comparison to the BioRad Bioplex 2200 series Syphilis Total (IgG/IgM), Wampole Impact RPR Test Kit, and to the Serodia Treponema pallidum particle agglutination assay (TP-PA).

The external clinical study along with in-house analytical studies will demonstrate the efficacy of the NOWDx Syphilis Test as an aid in the diagnosis of syphilis infection for at home testing and point of care testing sites. Participants will self test and be tested by Clinical Laboratory Improvement Amendments (CLIA) Waived operators with the NOWDx Syphilis Test at independent sites in WA, AZ, and NV. Two sample types will be tested with the NOWDx Syphilis Test for each participant: fingerstick whole blood and venous whole blood. Sera from each participant will be tested at an independent reference laboratory.

The NOWDx Syphilis Test will be evaluated in diverse populations of sexually active persons who self-select for syphilis testing and expectant mothers.

ELIGIBILITY:
* Sexually active persons who self-select for syphilis testing

  * n=840 participants; ~280 per study site
  * Inclusion criteria:

    - sexually active persons 18-64 years old
  * Exclusion criteria:

    * persons <18 years old; persons >64 years old;
    * persons with limited or no reading skills;
    * persons who previously participated in a NOWDx study
* Expectant mothers

  * n=222 participants; ~74 per study site
  * Inclusion criteria:

    - expectant mothers ≥18 years old
  * Exclusion criteria:

    * persons <18 years old;
    * persons with limited or no reading skills;
    * persons who previously participated in a NOWDx study
* Lay users

  * n=48 participants; ~16 per study site
  * Inclusion criteria:

    * persons 18-64 years old;
    * -½ high risk sexual behavior; ½ low risk sexual behavior
  * Exclusion criteria:

    * persons <18 years old; persons >64 years old;
    * persons with limited or no reading skills;
    * persons who previously participated in a NOWDx study

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Residents of the U.S. who elect to participate in the study
Sampling Method: Probability Sample
Enrollment: 1535 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Compare serological status to comparator method | through study completion, an average of 6 months
  The comparator method used in this study is an algorithm comprised of results from three different commercially available syphilis assays: an FDA-cleared treponemal immunoassay, an FDA-cleared non-treponemal assay (RPR assay) and a second treponemal assay (TP-PA).
Evaluate test reproducibility by lay users | through study completion, an average of 6 months
  Test lay user reproducibility using prepared samples for % agreement with expected results.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Rabine, MS, Study Director — NOW Diagnostics, Inc.
Locations (6):
- United States (6):
  - AMR Tempe, Tempe, Arizona
  - Matrix Clinical Research, Los Angeles, California
  - Segal Trials, North Miami, Florida
  - AMR Las Vegas, Las Vegas, Nevada
  - People Care Institute, West Orange, New Jersey
  - Multicare Rockwood, Cheney, Washington

IPD SHARING:
Plan to Share IPD: No